CLINICAL TRIAL: NCT01108692
Title: Investigation on Early Detection and Active Management of Supra-ventricular Arrhythmia With Telecardiology
Brief Title: Strategy of Early Detection and Active Management of Supraventricular Arrhythmia With Telecardiology (SETAM)
Acronym: SETAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik France (Industry)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS053
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Atrial Tachycardia
Keywords: atrial fibrillation; supraventricular arrhythmia; antithrombotic treatment; antiarrhythmic drugs; medical reaction time; telecardiology; early detection; holters memories; Pacemaker
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Blood Glucose Self-Monitoring; Remote Patient Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Patients will be followed by telecardiology.
  Interventions: Other: Telecardiology
- Control (Active Comparator): Patients will be followed in the conventional manner. They will be equipped with telecardiology but data will not be used for patient surveillance.
  Interventions: Other: Telecardiology

INTERVENTIONS:
Other: Telecardiology — Telecardiology will be switched on for both groups. For the Active group, all data will be transmitted to the physician. For the Control group, data will not be used for patients surveillance, only events regarding implant (Elective Replacement Indication) or events regarding data transmission missing will be generated and sent to the physician.
  A retrospective analysis will be performed at the end of the study to compare the results in the two groups.
  Other Names: Home-Monitoring; Remote monitoring

SUMMARY:
This study investigates if the early detection and treatment of supraventricular arrhythmia (SVA) may help to prevent the progression of the arrhythmia and improve the clinical outcome.

The primary endpoint investigates the delay to implement treatment in two groups of patients :

* Active group: Patients followed by telecardiology.
* Control group: Patients followed in the conventional manner.

It is assumed that the delay to implement treatment will be higher in the Control group.

DETAILED DESCRIPTION:
Atrial fibrillation is the most commonly encountered sustained cardiac arrhythmia in medical practice and it is often associated with atrial flutter. In patients with the new pacemaker generation EVIA, the home-monitoring technology provides specific and clinical relevant notifications for detection of atrial arrhythmias. Combined with holters memories, this can help to optimize the treatment of supraventricular arrhythmia (SVA) such as atrial fibrillation or flutter.

This study will compare in the two groups the delay to implement for the first time a treatment for the supraventricular arrhythmia (antiarrhythmic drugs and/or an antithrombotic treatment).

ELIGIBILITY:
Inclusion Criteria:

* Dual chamber pacemaker with activated Telecardiology
* CHAD2DS2-VASc score ≥ 2
* Sinusal rhythm at enrollment
* Patient willing and able to comply with the protocol
* Patient has provided informed consent
* Men and women > 18 years-old
* Patients geographically stable

Exclusion Criteria:

* Anticoagulation therapy
* Dual anti-platelet therapy
* Class I or class III anti-arrhythmic drugs
* Contraindication to antithrombotic therapy
* Participation in another clinical study
* Have a life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Delay to implement antithrombotic and/or antiarrhythmic drugs for the supraventricular arrhythmia. | 12-month
  Delay from enrollment until the next in-office follow-up during which the supraventricular arrhythmia is managed for the first-time.

SECONDARY OUTCOMES:
Serious adverse events related to supraventricular arrhythmia. | 12-month
  Including : Stroke, systemic embolic event, death, bleeding, and hospitalization for cardiac insufficiency
Atrial burden at the end of the study | 12-month
Atrial burden related to time | 12-month
  In order to check if atrial burden is time-dependent.
Supraventricular arrhythmia prevalence | 12-month
  Proportion of patients with supraventricular arrhythmia at the end of the 12-month follow-up.
Number of patients with managed supraventricular arrhythmia | 12-month
  Number of patients with supraventricular arrhythmia and for whom the physician implemented an overall management strategy (antithrombotic and/or antiarrhythmic drugs).
Supraventricular arrhythmia symptoms score (via a questionnaire) | at each follow-up visit
  Questionnaire submitted to the patient at enrollment and at each follow-up visit.
Quality of Life (via the EQ-5D Questionnaire) | at each follow-up visit
  The general health perception of the patients will be asked for, via the standardized EuroQOL EQ-5D questionnaire. This questionnaire provides a descriptive profile covering five dimensions (mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression) as well as a self-rating score of the patient's own assessment of its heath status.

CONTACTS AND LOCATIONS:
Overall Officials: Walid AMARA, MD, Principal Investigator — Intercommunal General Hospital in Montfermeil (93370 MONTFERMEIL- FRANCE)
Locations (57):
- France (57):
  - CH Général d'Abbeville, Abbeville
  - CH du Pays d'Aix, Aix-en-Provence
  - CH de la région d'Annecy, Annecy
  - CH d'Argentueil, Argenteuil
  - CH d'ARRAS, Arras
  - CH d'AURILLAC, Aurillac
  - CH d'AUXERRE, Auxerre
  - CH d'AVIGNON, Avignon
  - CH de Béziers, Béziers
  - CH de Blois, Blois
  - Centre Hospitalier Jacques Coeur, Bourges
  - Hôpital Sainte Camille, Bry-sur-Marne
  - CH de Cannes, Cannes
  - CH de Castres, Castres
  - CH William Morey, Chalon-sur-Saône
  - Les Hôpitaux de Chartres, Chartres
  - CH de CHATEAUROUX, Châteauroux
  - CH Public du Cotentin, Cherbourg
  - HIA Percy, Clamart
  - CHG Louis Pasteur, Colmar
  - Hôpital Schweitzer, Colmar
  - CH DINAN, Dinan
  - CH de DOLE, Dole
  - CH de DOUARNENEZ, Douarnenez
  - CHI Eure-Seine, Évreux
  - CH de Firminy, Firminy
  - CH d'HAGUENAU, Haguenau
  - CH de Jonzac, Jonzac
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - CH Saint Louis, La Rochelle
  - CH de Lagny, Lagny-sur-Marne
  - CH de LAVAL, Laval
  - CH A.Mignot, Le Chesnay
  - CH du Mans, Le Mans
  - CH de Lens, Lens
  - Groupe Hospitalier de l'Institut catholique de Lille, Lomme
  - CH de Longjumeau, Longjumeau
  - CH Bretagne Sud, Lorient
  - CHR Notre Dame de bon secours, Metz
  - CH de MONTAUBAN, Montauban
  - CH de MONTBELIARD, Montbéliard
  - CH Jean Bouveri, Montceau-les-Mines
  - Intercommunal General Hospital LE RAINCY- MONTFERMEIL, Montfermeil
  - CHR d'ORLEANS, Orléans
  - CH François Mitterand, Pau
  - CH de Roubaix, Roubaix
  - CH de SAINT BRIEUC, Saint-Brieuc
  - CHI du Val d'Ariège, Saint-Jean-de-Verges
  - CH de Saintonge, Saintes
  - CH de SAINT-MALO, St-Malo
  - CH Metz-Thionville Bel Air, Thionville
  - CH de TOULON, Toulon
  - CH de TROYES, Troyes
  - CH de Valence, Valence
  - CH de Valenciennes, Valenciennes
  - CH Bretagne Atlantique, Vannes
  - CHI de Villeneuve, Villeneuve-Saint-Georges